CLINICAL TRIAL: NCT04711655
Title: Double-blind, Placebo-controlled Clinical Trial on the Efficacy of Antireflux Ablation of the Cardiac Mucosa for the Treatment of Gastroesophageal Reflux Disease
Brief Title: Antireflux Ablation of the Cardia Mucosa vs Placebo for the Treatment of Gastroesophageal Reflux Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Collaborators: Spanish Society of Digestive Endoscopy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ECA-HRC-ARMA
Record Dates: First submitted 2020-12-21; First posted 2021-01-15 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2024-07

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: endoscopy; argon gas; antireflux ablation of the cardiac mucosa (ARMA)
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- (ARMA) antireflux ablation of the cardiac mucosa (Experimental): The ARMA (Ablation with electrocoagulation current or by argon gas fulguration) technique will be performed in patients assigned to this treatment arm.
  Interventions: Procedure: ARMA (antireflux ablation of the cardiac mucosa)
- upper digestive endoscopy (Placebo Comparator): Quality diagnostic upper gastrointestinal endoscopy will be performed without intervention in patients assigned to this treatment arm.
  Interventions: Procedure: upper digestive endoscopy

INTERVENTIONS:
Procedure: ARMA (antireflux ablation of the cardiac mucosa) — is an endoscopy in which argon gas ablation of the cardiac mucosa
  Arms: (ARMA) antireflux ablation of the cardiac mucosa
Procedure: upper digestive endoscopy — Quality diagnostic upper gastrointestinal endoscopy will be performed without intervention in patients assigned to this treatment arm.
  Arms: upper digestive endoscopy

SUMMARY:
The ARMA technique improves GORD-related quality of life with a low proportion of adverse effects.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is defined as the presence of symptoms or complications secondary to the passage of gastric contents into the esophagus, oral cavity or structures of the airway. The prevalence worldwide is between 8-33%. The clinical practice guidelines of the American College of Gastroenterology establish that first-line treatment, in the absence of alarm symptoms, should be carried out empirically. This treatment consists of hygienic-dietary measures and the use of proton pump inhibitors (PPIs) for 8-12 weeks. Despite the proven effectiveness of PPIs, there is 10-40% of patients who do not respond adequately to this treatment. All this has motivated the appearance of endoscopic and surgical techniques that offer an alternative to medical treatment. Among them is the technique of antireflux ablation of the cardiac mucosa (ARMA) in which the resection of the mucosa is replaced by an ablation with electrocoagulation current or by argon gas fulguration.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years.
2. GERD symptoms lasting more than 6 months, not necessarily consecutive. They should at least have a typical GERD symptom (heartburn or regurgitation).
3. Total acid exposure time> 6% in pH measurement study without PPI treatment.
4. Patients who do not want to take PPIs or with chronic consumption, defined as PPI consumption of more than 6 months (consecutive or not) in the last 2 years.
5. Response to PPI treatment, defined as an increase of> 10 points on the GERD-HRQL questionnaire 15 days after discontinuation of the PPI.
6. Written informed consent to participate in the study.

Exclusion Criteria:

1. Patients with sliding hiatal hernia> 2 cm.
2. Presence of only atypical GERD symptoms.
3. Age> 75 years.
4. Grade D peptic esophagitis.
5. Body mass index> 35 40 kg / m2.
6. Liver cirrhosis.
7. Pregnancy.
8. Incomplete relaxation of the LES in MAR (PIR> 15 mmHg).
9. Absent peristalsis, defined as 100% failed waves with DCI <100 mmHg * cm * s in MAR.
10. Esophagogastric surgery or previous endoscopic antireflux technique.
11. Barrett's esophagus with dysplasia.
12. Oncological disease.
13. Esophageal strictures or ulcers.
14. Severe cardiopulmonary comorbidity (ASA functional class IV-V).
15. Previously known coagulopathy.
16. Severe psychiatric disorder
17. Refusal to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the clinical efficacy (measured through the GERD-HRQL questionnaire) of the ARMA technique for the endoscopic treatment of PPI-dependent GERD. | The GERD-HRQL questionnaire score without PPI from visit 1 will be compared with the score without PPI from visit 4 (month 12).
  GERD-HRQL questionnaire score. Quantitative variable. Clinical success will be defined as a> 50% reduction in symptom score. The scale has 11 items. Each item is scored from 0 to 5, with a higher score indicating a better QOL.

SECONDARY OUTCOMES:
GERD-Q questionnaire score | The GERD-Q questionnaire score without PPI from visit 1 will be compared with the score without PPI from visit 4 (month 12).
  The GERDQ questionnaire is diagnostic for gastroesophageal reflux disease. Clinical success will be defined as a> 50% reduction in symptom score. The total Total score of 0 to 2 points = 0 % likelihood of GERD; 3 to 7 points = 50 %; 8 to 10 points = 79 %; 1 to 18 points = 89%;
PPI consumption | It is measured in the different visits after the intervention (month 1, month 3 and month 12)
  Ordinal qualitative variable: The patient will indicate if he feels satisfied / neutral / dissatisfied.
pHmetry-impedancemetry | This test will be performed on the patient before the intervention, in month 3 and in month 12
  Technique used to quantify acid, know when there is more acid reflux and correlate symptoms with the presence of that acid. one of the measurements that we are going to obtain with this test is acid exposure time.
High resolution manometry | This test will be performed on the patient before the intervention, in month 3 and in month 12
  This technique measures the pressure of esophageal contractions and with this technique different measurements are obtained such as lower esophageal sphincter resting pressure, integrated relaxation pressure, ICD.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique MD Rodríguez de Santiago, Principal Investigator — Servicio de Gastroenterología y Hepatología Hospital Ramón y Cajal
Locations (9):
- Spain (9):
  - Hospital de San Agustín, Avilés
  - Hospital Germans Trias I Pujol, Badalona
  - Hospital Del Mar, Barcelona
  - Hospital de Cabueñes, Gijón
  - Hospital 12 de Octubre, Madrid
  - Hospital La Paz, Madrid
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital La Fe, Valencia
  - Hospital Rio Hortega, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodriguez de Santiago E, Teruel Sanchez-Vegazo C, Albeniz E, Estremera-Arevalo F, Arrubla Gamboa A, Castel de Lucas I, Arribas Anta J, Marin-Gabriel JC, Diez Redondo P, Nunez Rodriguez H, Herreros de Tejada A, El Haira Martinez I, Riu Pons F, Naves J, Uchima H, Marin I, Duque Alcorta JM, Perez Corte D, De Maria P, Perez Enciso I, Garcia-Suarez C, Lorenzo-Zuniga V, Nogales O, Muriel A, Albillos A. Multicenter, double-blind, sham endoscopy-controlled, randomized trial evaluating the efficacy of anti-reflux mucosal ablation for the treatment of gastro-esophageal reflux disease. Endoscopy. 2025 Dec 31. doi: 10.1055/a-2780-0706. Online ahead of print. PMID 41475422